CLINICAL TRIAL: NCT02107092
Title: Open-label Extension to Study ZS-004 [Phase 3 Multicenter, Multi-phase, Multi-dose, Prospective, Randomized, Double-blind, Placebo-controlled Maintenance Study of Safety Efficacy of ZS (Sodium Zirconium Cycolsilicate) in Hyperkalemia.]
Brief Title: Open-label Safety & Efficacy of ZS (Sodium Zirconium Cyclosilicate)10g qd to Extend Study ZS-004 in Hyperkalemia.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ZS Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ZS-004E
Record Dates: First submitted 2014-04-03; First posted 2014-04-08 (Estimated); Results first posted 2018-08-15 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-07

CONDITIONS: Hyperkalemia
MeSH Terms: conditions — Hyperkalemia | interventions — sodium zirconium cyclosilicate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sodium Zirconium Cyclosilicate (Experimental): Open label oral administration of sodium zirconium cyclosilicate 10g once daily for 11 months.
  Interventions: Drug: Sodium Zirconium Cyclosilicate

INTERVENTIONS:
Drug: Sodium Zirconium Cyclosilicate — Oral 10g once daily with breakfast for 11 months.
  Other Names: ZS

SUMMARY:
Subjects who completed the Double-blind Randomized Maintenance Phase (DBRMP) Study Day 29 visit in ZS-004 (NCT 02088073) and have an i-STAT potassium value that is 3.5 to 6.2 mmol/l inclusive or who discontinued during ZS-004 due to hypo- or hyperkalemia in the DBRMP and have a mean i-STAT potassium value from two consecutive measurements at 0 and 60 minutes on Acute Phase Day 1/Maintenance Phase Day 1 that is 3.5 to 6.2 mmol/l inclusive may have the option to participate in ZS-004E (NCT 021070920). Subjects who discontinued from study ZS-004 due to any other reasons (e.g. adverse events, poor compliance, investigator decision) will not be entered into study ZS-004E. All subjects who continue into the extension study must begin dosing within two (2) days after the last dose of investigational product in ZS-004.

DETAILED DESCRIPTION:
All subjects with i-STAT potassium values between 3.5-5.5 mmol/l, inclusive at the ZS-004 (NCT 02088073) DBRMP Study Day 29 visit, who continue directly into the open-label extension study ZS-004E (NCT 021070920), will enter the Maintenance Phase (MP) and start on open-label ZS at a dose of 10g qd. All subjects with i-STAT potassium values > 5.5 mmol/l at the ZS-004 DBRMP Study Day 29 visit will undergo an acute treatment phase (AP) where they will receive ZS 10g three times a day (tid) for 24 (3 doses) or 48 hours (6 doses). If the subject's i-STAT potassium is between 3.5-5.0 mmol/l, inclusive after 24 (AP Study Day 2) or 48 hours (AP Study Day 3), the subject will enter the MP at a starting dose of 10g qd.

For subjects who discontinued during ZS-004 DBRMP due to hypo- or hyperkalemia baseline potassium values will be determined within 1 day of administration of the first dose in the ZS-004E extension study by taking two (2) consecutive i-STAT potassium measurements at 0 and 60 minutes (± 10 minutes). If the mean i-STAT value is between 3.5 - 5.5 mmol/l, inclusive, the subject will enter directly into the MP and receive 10g ZS qd; if the mean i-STAT potassium value is > 5.5 mmol/l, the subject will enter the AP. If i-STAT potassium values are still >5.0 mmol/l on the morning of AP Study Day 3, subjects will not enter the MP but will be referred to their normal health care provider for standard of care.

If the i-STAT potassium value increases above 5.5 mmol/l during the MP with treatment at 10g qd, the dose can be increased to15g qd. Conversely, if S-K decreases to between 3.0-3.4 mmol/l, inclusive, the dose of ZS can be decreased in 5g qd, decrements. If a subject is on a 5g qd dose and still develops blood potassium i-STAT values between 3.0 - 3.4mmol, inclusive the dose can be reduced to 5g every other day.

Subjects will receive up to 11 months of treatment with open-label ZS.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent.
* Completed the ZS-004 DBRMP Study Day 29 visit or discontinued study ZS-004 during the DBRMP due to hypo- or hyperkalemia and able to start dosing in ZS-004E within two (2) days after the last dose of Investigational product in ZS-004.
* Subject must have an i-STAT potassium value that is 3.5 to 6.2 mmol/l inclusive at the ZS-004 DBRMP Study Day 29 visit or a mean i-STAT potassium value from two consecutive measurements at 0 and 60 minutes on Acute Phase Day 1/Maintenance Phase Day 1 that is 3.5 to 6.2 mmol/l inclusive if the subject discontinued study ZS-004 during the DBRMP due to hypo- or hyperkalemia .

Exclusion Criteria:

* Pseudohyperkalemia signs and symptoms, such as excessive fist clenching hemolyzed blood specimen, history of severe leukocytosis or thrombocytosis.
* Subjects who received alternative treatment for hyperkalemia while participating in study ZS-004.
* Subjects with a life expectancy of less than 3 months.
* Subjects who are severely physically or mentally incapacitated and who in the opinion of investigator are unable to perform the subjects' tasks associated with the protocol.
* Women who are pregnant, lactating, or planning to become pregnant.
* Subjects with diabetic ketoacidosis.
* Presence of any condition which, in the opinion of the investigator, places the subject at undue risk or potentially jeopardizes the quality of the data to be generated.
* Known hypersensitivity or previous anaphylaxis to ZS or to components thereof.
* Treatment with a drug or device other than ZS within the last 30 days that has not received regulatory approval at the time of study entry.
* Subjects with cardiac arrhythmias that require immediate treatment.
* Subjects on dialysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2014-05-31 (Actual); Primary Completion 2015-07-31 (Actual); Study Completion 2015-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Rasmussen, MD, PhD, Study Chair — ZS Pharma, Inc.
Locations (46):
- United States (38):
  - Anniston, Alabama
  - Huntsville, Alabama
  - Scottsboro, Alabama
  - Phoenix, Arizona
  - Tempe, Arizona
  - Hawaiian Gardens, California
  - Los Angeles, California
  - Paramount, California
  - Riverside, California
  - Atlantis, Florida
  - Bradenton, Florida
  - Brandon, Florida
  - Brooksville, Florida
  - DeLand, Florida
  - Edgewater, Florida
  - Miami, Florida
  - Miami Lakes, Florida
  - New Smyrna Beach, Florida
  - Ocala, Florida
  - Summerfield, Florida
  - Tampa, Florida
  - Winter Park, Florida
  - Columbus, Georgia
  - Decatur, Georgia
  - Evergreen Park, Illinois
  - Joliet, Illinois
  - Shreveport, Louisiana
  - Auburn, Maine
  - Chesterfield, Michigan
  - Kansas City, Missouri
  - Las Vegas, Nevada
  - Flushing, New York
  - Altoona, Pennsylvania
  - Providence, Rhode Island
  - Orangeburg, South Carolina
  - Sumter, South Carolina
  - Chattanooga, Tennessee
  - San Antonio, Texas
- Australia (5):
  - Gosford, New South Wales
  - Woolloongabba, Queensland
  - Heidelberg, Victoria
  - Melbourne, Victoria
  - Parkville, Victoria
- South Africa (3):
  - Meyerspark
  - Port Elizabeth
  - Somerset West

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 30 outpatient sites in the United States, Australia and South Africa from 10 May 2014 to 14 July 2015.
Pre-assignment Details: Participants that completed Study ZS-004 (NCT02088073) Extended Dosing (ED) Phase Study Day 29 Visit or discontinued Study ZS-004 during the ED Phase due to hypo- or hyperkalemia, had a mean i-STAT potassium value between 3.5 and 6.2 mmol/L, and were able to start dosing in Study ZS-004E within 2 days after the last dose of study drug in ZS-004.
Groups:
- Extended Dosing Phase: ZS (Sodium Zirconium Cyclosilicate) QD: ZS 10g QD starting dose. ZS dose was increased or decreased in increments/ decrements of 5g QD to maximum of 15g QD or minimum of 5g every other day (QOD) if i-STAT potassium values increased to > 5.5 mmol/L or decreased to between 3.0 and 3.4 mmol/L, respectively.
Period: Overall Study
Arm/Group | Extended Dosing Phase: ZS (Sodium Zirconium Cyclosilicate) QD
Started | 123
Completed | 79
Not Completed | 44
Not completed — Miscellaneous | 3
Not completed — Subject compliance | 3
Not completed — Hypo-or hyperkalemia | 2
Not completed — Met ECG withdrawal criteria | 3
Not completed — Physician Decision | 3
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 9
Not completed — Adverse Event | 7
Not completed — Expected progression of CKD | 12

BASELINE CHARACTERISTICS:
Population: 2 subjects did not have any S-K measurements during the ED phase due to early termination and are excluded from baseline characteristics
Arm/Group | Extended Dosing Phase: ZS (Sodium Zirconium Cyclosilicate) QD
Number analyzed (Participants) | 121
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.7 (12.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 70
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2
  Black or African American | 11
  White | 107
  Other | 1
Study ZS-004 Acute Phase S-K baseline [Count of Participants; unit: Participants] — Acute Phase S-K baseline of participants in Study ZS-004
  Participants
    < 5.5 mmol/L | 54
    5.5-< 6.0 mmol/L | 53
    ≥ 6.0 mmol/L | 14
Acute Phase eGFR at baseline [Count of Participants; unit: Participants] — Acute Phase baseline from Study ZS-004
  Participants
    <60 mL/min | 90
    ≥ 60 mL/min | 31
Cormordid conditions and concomitant medications which may contirubute to hyperkalemia [Number; unit: Participants] — Categories are not mutually exclusive
  Participants
    RAAS inhibitor medication | 83
    Diabetes mellitus | 80
    Chronic kidney disease | 76
    Heart failure | 50

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects With Average Serum Potassium Values ≤ 5.1 mmol/L
Description: The proportions of subjects with average serum potassium (S-K) values ≤ 5.1 mmol/L during Extended Dosing Study Days 8 to 337, inclusive
Time Frame: 11 months
Population: Entered Extended Dosing Phase, received study drug and had post baseline S-K values during the Extended Dosing Phase. The analysis population includes 121 subjects, where there is one subject who only had end-of-study post-baseline measurement and therefore was not presented in the participants analyzed.
Measure: Number (95% Confidence Interval); unit: Proportion of Participants
Arm/Group | Extended Dosing Phase: ZS (Sodium Zirconium Cyclosilicate) QD
Number analyzed (Participants) | 120
Proportion of Participants
  ED Study Day 8 | 0.875 [0.802 to 0.928]
  ED Study Day 15: number analyzed (Participants) | 118
  ED Study Day 15 | 0.822 [0.741 to 0.886]
  ED Study Day 22: number analyzed (Participants) | 118
  ED Study Day 22 | 0.797 [0.713 to 0.865]
  ED Study Day 29: number analyzed (Participants) | 116
  ED Study Day 29 | 0.862 [0.786 to 0.919]
  ED Study Day 36: number analyzed (Participants) | 112
  ED Study Day 36 | 0.848 [0.768 to 0.909]
  ED Study Day 43: number analyzed (Participants) | 111
  ED Study Day 43 | 0.793 [0.705 to 0.864]
  ED Study Day 50: number analyzed (Participants) | 108
  ED Study Day 50 | 0.796 [0.708 to 0.868]
  ED Study Day 57: number analyzed (Participants) | 107
  ED Study Day 57 | 0.766 [0.675 to 0.843]
  ED Study Day 85: number analyzed (Participants) | 88
  ED Study Day 85 | 0.807 [0.709 to 0.833]
  ED Study Day 113: number analyzed (Participants) | 84
  ED Study Day 113 | 0.798 [0.696 to 0.877]
  ED Study Day 141: number analyzed (Participants) | 81
  ED Study Day 141 | 0.815 [0.713 to 0.892]
  ED Study Day 169: number analyzed (Participants) | 70
  ED Study Day 169 | 0.771 [0.656 to 0.863]
  ED Study Day 197: number analyzed (Participants) | 68
  ED Study Day 197 | 0.809 [0.695 to 0.894]
  ED Day Study 225: number analyzed (Participants) | 65
  ED Day Study 225 | 0.846 [0.735 to 0.924]
  ED Study Day 253: number analyzed (Participants) | 63
  ED Study Day 253 | 0.778 [0.655 to 0.873]
  ED Study Day 281: number analyzed (Participants) | 60
  ED Study Day 281 | 0.833 [0.715 to 0.917]
  ED Study Day 309: number analyzed (Participants) | 58
  ED Study Day 309 | 0.828 [0.706 to 0.914]
  ED Study Day 337: number analyzed (Participants) | 51
  ED Study Day 337 | 0.843 [0.714 to 0.930]
  ED Study Day 337/Exit | 0.783 [0.699 to 0.853]
  ED Study Days 8-337 Average | 0.883 [0.812 to 0.935]

2. Secondary Outcome: Proportion of Subjects With Average Serum Potassium Values ≤ 5.5 mmol/L
Description: The proportions of subjects with average S-K values ≤ 5.5 mmol/L during Extended Dosing Study Days 8 to 337, inclusive
Time Frame: 11 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Proportion of Participants
Arm/Group | Extended Dosing Phase: ZS (Sodium Zirconium Cyclosilicate) QD
Number analyzed (Participants) | 120
Proportion of Participants
  ED Study Day 8 | 0.950 [0.894 to 0.981]
  ED Study Day 15: number analyzed (Participants) | 118
  ED Study Day 15 | 0.932 [0.871 to 0.970]
  ED Study Day 22: number analyzed (Participants) | 118
  ED Study Day 22 | 0.975 [0.927 to 0.995]
  ED Study Day 29: number analyzed (Participants) | 116
  ED Study Day 29 | 0.957 [0.902 to 0.986]
  ED Study Day 36: number analyzed (Participants) | 112
  ED Study Day 36 | 0.955 [0.899 to 0.985]
  ED Study Day 43: number analyzed (Participants) | 111
  ED Study Day 43 | 0.946 [0.886 to 0.980]
  ED Study Day 50: number analyzed (Participants) | 108
  ED Study Day 50 | 0.935 [0.871 to 0.974]
  ED Study Day 57: number analyzed (Participants) | 107
  ED Study Day 57 | 0.944 [0.882 to 0.979]
  ED Study Day 85: number analyzed (Participants) | 88
  ED Study Day 85 | 0.943 [0.872 to 0.981]
  ED Study Day 113: number analyzed (Participants) | 84
  ED Study Day 113 | 0.940 [0.867 to 0.980]
  ED Study Day 141: number analyzed (Participants) | 81
  ED Study Day 141 | 0.938 [0.862 to 0.980]
  ED Study Day 169: number analyzed (Participants) | 70
  ED Study Day 169 | 0.929 [0.841 to 0.976]
  ED Study Day 197: number analyzed (Participants) | 68
  ED Study Day 197 | 0.941 [0.856 to 0.984]
  ED Day Study 225: number analyzed (Participants) | 65
  ED Day Study 225 | 0.985 [0.917 to 1.000]
  ED Study Day 253: number analyzed (Participants) | 63
  ED Study Day 253 | 0.937 [0.845 to 0.982]
  ED Study Day 281: number analyzed (Participants) | 60
  ED Study Day 281 | 0.950 [0.861 to 0.990]
  ED Study Day 309: number analyzed (Participants) | 58
  ED Study Day 309 | 0.914 [0.810 to 0.971]
  ED Study Day 337: number analyzed (Participants) | 51
  ED Study Day 337 | 0.980 [0.896 to 1.000]
  ED Study Day 337/Exit | 0.942 [0.884 to 0.976]
  ED Study Days 8-337 Average | 1.000 [0.970 to 1.000]

ADVERSE EVENTS:
Time Frame: Eleven months
Description: The Extended Dosing Phase Safety Population was defined as all subjects who received at least 1 Extended Dosing Phase dose administration with any post-baseline Extended Dosing Phase safety data.
Groups:
- ZS (Sodium Zirconium Cyclosilicate) QD Extended Phase Dosing: ZS 10g QD starting dose increased or decreased in increments/ decrements of 5g QD to maximum of 15g QD or minimum of 5g QOD if i-STAT potassium values increased to > 5.5 mmol/L or decreased to between 3.0 and 3.4 mmol/L, respectively.
Arm/Group | ZS (Sodium Zirconium Cyclosilicate) QD Extended Phase Dosing
Serious Adverse Events (participants affected / at risk) | 24/123
Other Adverse Events (participants affected / at risk) | 82/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ZS (Sodium Zirconium Cyclosilicate) QD Extended Phase Dosing (N=123)
Anaemia (Blood and lymphatic system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 2
Myocardial infarction (Cardiac disorders) | 1
Retinal artery occlusion (Eye disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 2
Gastritis haemorrhagic (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Diabetic foot infection (Infections and infestations) | 1
Gangrene (Infections and infestations) | 1
Lobar pneumonia (Infections and infestations) | 1
Localised infection (Infections and infestations) | 1
Morganella infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Sepsis (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
Patella fracture (Injury, poisoning and procedural complications) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Dry gangrene (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ZS (Sodium Zirconium Cyclosilicate) QD Extended Phase Dosing (N=123)
Anaemia (Blood and lymphatic system disorders) | 6
Cardiac failure (Cardiac disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 7
Diarrhoea (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 4
Oedema (General disorders) | 4
Oedema peripheral (General disorders) | 10
Seasonal allergy (Immune system disorders) | 3
Gastroenteritis (Infections and infestations) | 3
Influenza (Infections and infestations) | 3
Pneumonia (Infections and infestations) | 3
Upper respiratory tract infection (Infections and infestations) | 5
Urinary tract infection (Infections and infestations) | 11
Blood urea increased (Investigations) | 3
Gout (Metabolism and nutrition disorders) | 4
Hyperlipidemia (Metabolism and nutrition disorders) | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6
Dizzines (Nervous system disorders) | 3
Headache (Nervous system disorders) | 4
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Hypertension (Vascular disorders) | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
ZS Pharma has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome. The PIs also agree for data to be presented first as a joint, multi-center publication.